CLINICAL TRIAL: NCT06451627
Title: Esketamine on Postoperative Sleep Disturbance of Patients Undergoing Spinal Surgery：A Randomized Controlled Trial
Brief Title: Esketamine on Postoperative Sleep Disturbance of Patients Undergoing Spinal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ruquan Han, Director, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: esketamine-JMY
Record Dates: First submitted 2024-05-11; First posted 2024-06-11 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-06

CONDITIONS: Esketamine; Sleep Disturbance; Spinal Surgery
MeSH Terms: conditions — Parasomnias | interventions — Esketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- esketamine (Experimental): Esketamine ( 50mg, dissolved in 50ml normal saline ) will be infused at a speed of 0.3mg / kg / h during surgery .Total intravenous anesthesia with propofol ,remifentanil will be implemented for anesthesia maintenance based on the bispectral index(BIS) and keep BIS between 40-60 .
  Interventions: Drug: Esketamine
- saline (Placebo Comparator): Saline will be infused at a speed of 0.3mg / kg / h during surgery .Total intravenous anesthesia with propofol ,remifentanil will be implemented for anesthesia maintenance based on the bispectral index(BIS) and keep BIS between 40-60 .
  Interventions: Drug: saline

INTERVENTIONS:
Drug: Esketamine — Esketamine ( 50mg, dissolved in 50ml normal saline ) will be infused at a speed of 0.3mg / kg / h during surgery .
  Arms: esketamine
Drug: saline — Saline will be infused at a speed of 0.3mg / kg / h during surgery .
  Arms: saline

SUMMARY:
The goal of this clinical trial is to learn about the effect of intraoperative esketamine infusion on postoperative sleep disturbance(PSD) of patients undergoing spinal surgery. The main aims to answer are:

* To explore the effect of intraoperative infusion of esketamine on the incidence of postoperative sleep disturbance and sleep quality in patients undergoing spinal surgery.
* To explore the effect of intraoperative infusion of esketamine on postoperative pain, anxiety and depression ; Participants will be patients undergoing spinal surgery with general anesthesia at Beijing Tiantan Hospital. 0.3mg/kg/h esketamine or saline will be infused during surgery . The incidence of sleep disturbance , sleep quality, pain scores, hospital anxiety and depression scores and perioperative adverse events after surgery will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old,
* American Society of Anesthesiologist (ASA) Physical Status classification I to III ;
* Patients scheduled to undergo elective spinal surgery under general anesthesia;
* Signed informed consent ;

Exclusion Criteria:

* BMI > 35kg / m2 ;
* Severe lesions of important organs and systems ;
* The estimated duration of surgery is more than 4 hours
* Patients who were retained tracheal intubation or admitted to intensive care unit (ICU) postoperatively.
* History of adverse reactions or contraindications to ketamine and esketamine ;
* Cognitive dysfunction, communication disorders ;
* Refused to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2025-12-28 (Estimated); Study Completion 2026-01-28 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative sleep disturbance(PSD) in patients undergoing spinal surgery | during the first three days after surgery
  It will be evaluated by Athens Insomnia Scale (AIS) on the morning(8-10 am) of postoperative days 1-3, a score of 6 or higher will be defined as PSD.

SECONDARY OUTCOMES:
objective sleep quality(total sleep time) of patients with spinal surgery assesssed by the sleep monitoring equipment. | on the postoperative day 1 and postoperative day 3 after surgery
  It will be evaluated by an sleep monitoring equipment which can record total sleep time in hour.
The pain scores | within 72hours after surgery
  Postoperative pain at rest and movement will be evaluated on the morning(8-10 am) of postoperative days 1-3 using NRS.0 indicating no pain, 10 indicating worst pain imaginable.
dosage of analgesics | within 72 hours after surgery
  The analgesic consumption(PCIA) and supplemental analgesics within 72h will be recorded.
Postoperative hospital anxiety and depression scale ( HADS ) score. | on the postoperative day 1 and postoperative day 3 after surgery
  Postoperative anxiety and depression scores will be measured by the Hospital Anxiety and Depression Scale, on the morning(8-10 am) of postoperative days (PODs) 1 and 3 , a score of 8 points or higher will be diagnosed as depression or anxiety.

OTHER OUTCOMES:
The incidence of all drug-related adverse events | within 72hours after surgery
  All drug-related adverse events including bradycardia, hypotension, tachycardia, hypertension, arrhythmia, nystagmus, hypersalivation, euphoria, emergence agitation, hallucinations, dreaminess and nightmares during surgery or before discharge.etc.Patients will be followed up for 3 days consecutively(at 8-10am).

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tian Tan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
All data generated or analysed during this study will be included in published article. The data that support the findings of this study are available from the corresponding author, HW upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Access Criteria: The data that support the findings of this study are available from the corresponding author, HW upon reasonable request.

REFERENCES:
- [Derived] Jian M, Chen Y, Wang S, Zhou Y, Liu H, Liang F, Han R, Wang H. Effect of esketamine on postoperative sleep disturbance in patients undergoing spinal surgery: a study protocol for a randomised, double-blinded, placebo-controlled clinical trial. BMJ Open. 2025 Mar 4;15(3):e090089. doi: 10.1136/bmjopen-2024-090089. PMID 40037679